CLINICAL TRIAL: NCT01051596
Title: A Phase II Study of ABT-888, an Inhibitor of Poly(ADP-ribose) Polymerase (PARP) in Combination With Temozolomide in Patients With Heavily Pretreated, Metastatic Colorectal Cancer
Brief Title: A Study of ABT-888 in Combination With Temozolomide for Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Michael J Pishvaian, Assistant Professor of Medicine, Georgetown University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-170
Record Dates: First submitted 2010-01-08; First posted 2010-01-18 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Cancer
Keywords: metastatic; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Temozolomide; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ABT-888 and temozolomide (Experimental): Temozolomide Days 1-5 and ABT-888 Days 1-7 of each 28-day cycle
  Interventions: Drug: Temozolomide; Drug: ABT-888

INTERVENTIONS:
Drug: Temozolomide — 150mg/m2 Days 1-5 of each 28 day cycle
  Other Names: Temodar
Drug: ABT-888 — 40mg orally BID Days 1-7 of each 28 day cycle
  Other Names: Veliparib

SUMMARY:
People with colorectal cancer that cannot be cured by surgery are being asked to participate in this study.

The purpose of this study is to test the efficacy (effectiveness) of a new combination of drugs, ABT-888 and temozolomide for patients with colorectal cancer. Temozolomide acts by damaging deoxyribonucleic acid (DNA) in rapidly dividing cells, in other words, cancer cells. ABT-888 inhibits an enzyme called "PARP" which helps to fix damaged DNA. By inhibiting this enzyme, ABT-888 prevents cancer cells from repairing the damage caused by the temozolomide, and will hopefully increase the killing of cancer cells, and decrease the tumors in the body.

ABT-888 is an investigational or experimental anti-cancer agent that has not yet been approved by the Food and Drug Administration (FDA) for use in colorectal cancer.

This study will help find out what effects (good and bad) the combination of drugs, temozolomide and ABT-888 has on colorectal cancer.

This research is being done because it is not known if ABT-888 will increase the effectiveness of temozolomide for colorectal cancer.

DETAILED DESCRIPTION:
We will initiate a single arm, open label Phase II study to test the clinical activity of ABT-888 and temozolomide in patients with metastatic colorectal cancer.

Treatment will continue weekly with restaging scans to be performed every 8 weeks. The trial will follow a Simon's two-stage optimal design. For the first stage, 21 patients will be accrued. If two (9.5%) or fewer of the 21 patients exhibit a partial or complete response with ABT-888 plus temozolomide, the agent will be rejected and the trial stopped. However, if at least 3 patients of the 21 (14%) exhibit a response in the first stage, then an additional 29 patients will be entered into the second stage, for a total of 50 patients in this phase II study. If 8 (16%) or more patients exhibit a response, then the treatment will be considered for further investigation. The sample sizes of 21 and 50 patients and the decision rules, in stages 1 and 2 respectively, are designed to differentiate a 25% overall response rate from a 10% overall response rate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven colorectal cancer with measurable or evaluable disease
* Progression on or intolerance of or ineligibility for all standard therapies (including regimens containing fluoropyrimidine, oxaliplatin, irinotecan, bevacizumab, and an anti-EGFR antibody (where appropriate))
* Age > = 18 years
* ECOG performance status 0-2
* Subjects with no brain metastases or a history of previously treated brain metastases who have been treated by surgery or stereotactic radiosurgery at least 4 weeks prior to enrollment and have a baseline MRI that shows no evidence of active intercranial disease and have not had treatment with steroids within 1 week of study enrollment
* At least 21 days since prior anti-cancer therapy, including chemotherapy, biological therapy, radiation therapy or any investigational agent within 4 weeks before starting ABT-888 and temozolomide
* Adequate hepatic, bone marrow, and renal function
* Partial thromboplastin time (PTT) must be </= 1.5 x the upper limit of institution's normal range and INR < 1.5. Subjects on anticoagulant will have PTT and INR as determined by the investigator.
* Subject's with significant fluid retention, including ascites or pleural effusion, may be allowed at the discretion of the PI
* Life expectancy > 12 weeks
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to initiation of treatment and/or postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Subject is capable of understanding and complying with parameters as outlined in the protocol and able to sign and date the informed consent approved by the IRB prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

* CNS metastases which do not meet the criteria outlined in inclusion criteria
* Active severe infection or known chronic infection with HIV, hepatitis B virus, or hepatitis C virus
* Cardiovascular disease problems including unstable angina, therapy for life-threatening ventricular arrhythmia, myocardial infarction, stroke or congestive heart failure within the last 6 months
* Life threatening visceral disease or other severe concurrent disease
* Women who are pregnant or breastfeeding
* Anticipated patient survival under 3 months
* The subject has had another active malignancy within the past five years except for cervical cancer in site, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin.
* Clinically significant and uncontrolled major medical conditions including but not limited to: active uncontrolled infection, symptomatic congestive heart failure, Unstable angina pectoris or cardiac arrhythmia, psychiatric illness/ social situation that would limit compliance with study requirements; any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-09; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Pishvaian, MD, PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Pishvaian MJ, Slack RS, Jiang W, He AR, Hwang JJ, Hankin A, Dorsch-Vogel K, Kukadiya D, Weiner LM, Marshall JL, Brody JR. A phase 2 study of the PARP inhibitor veliparib plus temozolomide in patients with heavily pretreated metastatic colorectal cancer. Cancer. 2018 Jun 1;124(11):2337-2346. doi: 10.1002/cncr.31309. Epub 2018 Mar 26. PMID 29579325

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABT-888 and Temozolomide
Started | 75
Completed | 75
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ABT-888 and Temozolomide
Number analyzed (Participants) | 75
Age, Continuous [Median (Full Range); unit: years] | 56 [35 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 48
  More than one race | 0
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With Disease Control
Description: Disease control rate defined as stable disease, partial response, or complete response according to the Response Evaluation Criteria in Solid Tumors (RECIST).
Time Frame: 2 months
Population: Percent of patients with disease control, according to the Response Evaluation Criteria in Solid Tumors (RECIST).
Measure: Count of Participants; unit: Participants
Arm/Group | ABT-888 and Temozolomide
Number analyzed (Participants) | 75
Participants | 18

2. Secondary Outcome: Median Progression-free Survival Time
Description: Progression-free survival defines as the time in days from study study entry until progression or death
Time Frame: 1 year
Population: All patients were evaluable for response, on an intention to treat basis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ABT-888 and Temozolomide
Number analyzed (Participants) | 75
Months | 1.8 [1.6 to 1.9]

3. Secondary Outcome: Overall Survival
Description: Overall survival defined as the time in days from study entry until death
Time Frame: 1 year
Population: All patients were evaluable for response, on an intention to treat basis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ABT-888 and Temozolomide
Number analyzed (Participants) | 75
Months | 6.6 [5.6 to 7.4]

4. Secondary Outcome: Percent of Patients With an Objective Response
Description: Objective response rate defined as partial response or complete response according to RECIST criteria
Time Frame: 2 months
Population: All patients were evaluable for response, on an intention to treat basis
Measure: Count of Participants; unit: Participants
Arm/Group | ABT-888 and Temozolomide
Number analyzed (Participants) | 75
Participants | 2

ADVERSE EVENTS:
Arm/Group | ABT-888 and Temozolomide
Serious Adverse Events (participants affected / at risk) | 5/75
Other Adverse Events (participants affected / at risk) | 75/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABT-888 and Temozolomide (N=75)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — Fevers and low neutrophil count
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) — Low platelets
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABT-888 and Temozolomide (N=75)
Thrombocytopenia (Blood and lymphatic system disorders) | 40 — Low Platelets
Anemia (Blood and lymphatic system disorders) | 35 — Low red blood cells
Leucopenia (Blood and lymphatic system disorders) | 15 — Low white blood cells
Neutropenia (Blood and lymphatic system disorders) | 13 — Low neutrophils
Lymphopenia (Blood and lymphatic system disorders) | 2 — Low lymphocytes
Fatigue (General disorders) | 19
Fever (General disorders) | 2
Weight loss (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Peeling of feet (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 36
Vomiting (Gastrointestinal disorders) | 14
Anorexia (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dysgeusia (Gastrointestinal disorders) | 1
Urinary Hemorrhage (Blood and lymphatic system disorders) | 1
Vaginal hemorrhage (Blood and lymphatic system disorders) | 1
Petechiae/Purpura (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Infections and infestations) | 1
Edema: limb (Blood and lymphatic system disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Elevated creatinine (Metabolism and nutrition disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 2
Pain NOS (General disorders) | 3
Headache (Nervous system disorders) | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes